CLINICAL TRIAL: NCT06229197
Title: Billroth II With Braun Anastomosis Versus Billroth II Anastomosis After Radical Distal Gastrectomy With D2 Lymphadenectomy for Gastric Cancer: a Randomized Controlled Trial
Brief Title: Billroth II With Braun Anastomosis After Radical Distal Gastrectomy for Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Bo Zhang, MD, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023HXFH005
Record Dates: First submitted 2024-01-01; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Surgery; Anastomosis; Gastrostomy
Keywords: Gastric Cancer; Gastrostomy; Billroth II; Braun Anastomosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Billroth II with Braun Reconstruction (Experimental)
  Interventions: Procedure: Billroth II reconstruction; Procedure: Braun Anastomosis
- Billroth II Reconstruction (Active Comparator)
  Interventions: Procedure: Billroth II reconstruction

INTERVENTIONS:
Procedure: Billroth II reconstruction — Billroth II reconstruction, in which a loop of jejunum is mobilized and anastomosed to the gastric remnant
Procedure: Braun Anastomosis — This is an additional surgical connection (anastomosis) created between two parts of the small intestine, specifically between the afferent (incoming) and efferent (outgoing) limbs of the jejunum near the gastrojejunostomy (the new connection between the stomach and small intestine created during a Billroth II procedure).
  Arms: Billroth II with Braun Reconstruction

SUMMARY:
The primary aim of this trial is to rigorously evaluate the comparative benefits and potential risks associated with Billroth II reconstruction with Braun anastomosis versus Billroth II reconstruction alone following distal gastrectomy with D2 lymphadenectomy in patients diagnosed with gastric cancer. This assessment focuses on delineating the therapeutic efficacy, safety profile, and overall clinical outcomes of these two surgical approaches in treating this condition.

ELIGIBILITY:
Inclusion criteria

To be enrolled, participants must be phase I-III patients with initial treatment of radical distal gastrectomy and satisfying the following inclusion criteria:

1. Histologically proven stage I-III gastric cancer, evaluated as radically resectable
2. No synchronous or metachronous cancers
3. Patients have signed informed consent forms
4. Age 18-80 years old
5. No malfunction of cardio-pulmonary, liver, and kidney, ECOG score 0-1
6. No emergency surgery needed

Exclusion criteria

Patients will be excluded according to the following criteria:

1. Pregnant or lactating women
2. Distant metastasis to the liver, lung, bone, supraclavicular lymph nodes, pelvic, or ovarian species and peritoneal dissemination
3. Ascites or cachexia
4. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, poorly controlled hypertension or diabetes
5. Participation in other clinical trials 4 weeks before the enrollment of this trial or still participating in other trials
6. Mental illness
7. Surgical history whose influence has not been eliminated
8. History of another gastric or esophageal malignancy, including stromal tumor, sarcoma, lymphoma, and carcinoid
9. Active infection with a fever of over 38°C
10. Poor compliance
11. Not suitable for this trial because of other clinical or laboratory conditions determined by the researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of reflux gastritis assessed according to RGB classification | 6 months, 12 months
  by endoscopic evaluation

SECONDARY OUTCOMES:
Quality of life assessed by the PGSAS-45 Scale | 6 months, 12 months
  The preoperative and postoperative QoL of patients between the two groups.
Nutritional status | 6 months, 12 months
  Changes in body weight (kg) or BMI from baseline
Time to first passage of flatus/stool | within 30 days after surgery
  Time taken to pass first stool or flatus
Postoperative complications (assessed according to the Clavien-Dindo) | within 30 days after surgery
  e.g., anastomotic leakage, anastomotic bleeding assessed by laboratory test in combination with clinical features, radiological diagnostic methods, endoscopy, diagnostic laparoscopy.
Long-term complications | 6 months, 12 months
  e.g., food residue and bile reflux (assessed according to the RGB classification).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhang, MD, Study Chair — Gastric Cancer Center, Department of General Surgery, West China Hospital, Sichuan University; Zhaolun Cai, MD, PhD, Principal Investigator — Gastric Cancer Center, Department of General Surgery, West China Hospital, Sichuan University